CLINICAL TRIAL: NCT00402259
Title: A Randomised, Double-Blind, Double-Dummy, Active-Controlled, Multicenter Study to Assess the Efficacy and Safety of Esomeprazole or Omeprazole for 5 Days in Subjects With Acute Non-Variceal Upper Gastrointestinal Bleeding
Brief Title: Efficacy and Safety Study of Esomeprazole vs Omeprazole to Treat Acute Non-Variceal Upper Gastrointestinal Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D961DL00004; Nexium PUB
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: acute non-variceal upper gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

INTERVENTIONS:
Drug: Esomeprazole IV
Drug: Omeprazole IV

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Esomeprazole and Omeprazole intravenous every 12 hours for 5 days in subjects with acute non-variceal upper gastrointestinal bleeding

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years.
* GI bleeding or with such signs within 48 hours as judged by the investigator as to have non-variceal upper GI bleeding.
* One endoscopically confirmed bleeding peptic ulcer or erosive gastritis

Exclusion Criteria:

* GI bleeding caused by Esophageal varices
* Mallory Weiss syndrome
* Zollinger-Ellison syndrome
* Suspicion of gastric malignancy at baseline endoscopy
* Post-Billroth-resection
* Unknown source of GI bleeding · 2.Unstable vital signs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2006-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy by assessment of proportion of subjects who present with no clinically significant bleeding after 5 days treatment

SECONDARY OUTCOMES:
Proportion of subjects who present with no clinically significant upper GI bleeding after 72-hour treatment
Time to absence of clinically significant upper GI bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca
Locations (7):
- China (7):
  - Research site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Xi’an, Shanxi
  - Research Site, Beijing
  - Research Site, Shanghai
  - Research Site, Tianjin